CLINICAL TRIAL: NCT06346132
Title: Effect of Virtual Reality on Patient's Comfort During Cardiac Electronic Device Implantation: a Randomized, Controlled Trial.
Brief Title: Effect of Virtual Reality on Patient's Comfort During Cardiac Electronic Device Implantation.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Schlotterbeck Hervé (Other)
Responsible Party: Sponsor-Investigator, Schlotterbeck Hervé, Principal Investigator, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-00043 CE 4516
Record Dates: First submitted 2024-03-12; First posted 2024-04-03 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Virtual Reality; Medical Device; Local Anesthesia; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): In this group, virtual reality will be added to usual care
  Interventions: Device: Virtual reality application
- Standard Group (No Intervention): In this group, no extra intervention will be added to usual care

INTERVENTIONS:
Device: Virtual reality application — In this group, virtual reality will be added to usual care
  Arms: Experimental Group

SUMMARY:
The purpose of this study is to assess the effect on patient's comfort of a virtual reality experience during a procedure of cardiac electronic device implantation under local anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 year old,
* Patients who signed the consent form and accepted to participate to the trial,
* New cardiac electronic device implantation or cardiac electronic device battery change,
* Surgical procedure planned in ambulatory care.

Exclusion Criteria:

* Communication limitations,
* Surgical procedure planned in sedation or narcosis,
* Severe sensorial deficits (visual, auditory),
* Claustrophobia,
* Known motion sickness,
* Patient isolated or with contact precautions,
* Known or anticipated psychiatric diseases,
* Patient known for epilepsia,
* Opened scar and or ongoing infection at the level of the face and/or eyes,
* Patient evaluated non suitable for the study by the surgeon, cardiologist or anesthetist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Global pain intensity experienced during the procedure. | At the end of surgery
  Global pain intensity experienced during the procedure evaluated with the Visual Analogue Scale (VAS).

SECONDARY OUTCOMES:
Need for supplementary sedation and/or analgesia during the procedure. | At the end of surgery
  The need for supplementary sedation and/or analgesia during the procedure will be recorded. The doses of the drugs will be recorded.
Global anxiety intensity experienced during the procedure. | At the end of surgery
  Global anxiety intensity experienced during the procedure evaluated with the Visual Analogue Scale (VAS).
Patient's comfort during the procedure assessed by the surgeon and cardiologist. | At the end of surgery
  Patient's comfort during the procedure assessed by the surgeon and cardiologist using the Numeric Rating Scale (NRS).
Incidence of motion sickness during the virtual reality experience. | At patient discharge (or at a maximum of 4 hours after the end of surgery)
  Incidence of motion sickness during the virtual reality experience (for example nausea)
Patient's perceived procedure duration. | At the end of surgery
  Patient's perceived procedure duration compared to effective procedure duration.
Maximal systolic arterial blood pressure. | At the end of surgery
  Maximal systolic arterial blood pressure recorded during the procedure.
Incidence of hypotensive or hypoxic events during procedure. | At the end of surgery
  Incidence of hypotensive events (defined by systolic arterial blood pressure less than 90 mmhg) and/or hypoxic events (defined by oxygen saturation under 90%) during the procedure.
Total dose of local anaesthetic used during the procedure. | At the end of surgery
  Total dose of local anaesthetic used during the procedure (total dose in mg).
Change in anesthetic strategy during procedure. | At the end of surgery
  If a change of anesthesiologic strategy is needed during the procedure (for example, if the patient needs an unplanned general anesthesia during the procedure).
Interruption of virtual reality experience during the procedure. | At the end of surgery
  If the patient choose to remove the virtual reality headset and interrupt the virtual reality experience during the procedure.
Intra- and post-procedure complications. | At patient discharge (or at a maximum of 4 hours after the end of surgery)
  Registration of any complication during and after the procedure.
Overall patient's comfort and satisfaction experienced during the procedure. | At patient discharge (or at a maximum of 4 hours after the end of surgery)
  Overall patient's comfort and satisfaction experienced during the procedure assessed with Likert's scale (5 points).

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto CardioCentro, Lugano, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No